CLINICAL TRIAL: NCT03621332
Title: The HOLISTIC Study: Health-related Quality Of Life in Patients With Advanced Soft Tissue Sarcomas Treated With Chemotherapy
Brief Title: HRQoL in Advanced Soft Tissue Sarcoma Patients Treated With Chemotherapy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4782
Record Dates: First submitted 2018-07-19; First posted 2018-08-08 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Quality of Life
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire adminstration: All patients who participate will complete questionnaires
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Online/paper questionnaires

SUMMARY:
The benefits of cancer treatments, such as chemotherapy, are traditionally measured by outcomes such as progression free survival and overall survival. The degree to which treatments affect symptoms of disease, patient functioning and HRQoL are rarely measured or incorporated in the main endpoints of large-scale clinical trials. Systemic treatments for the majority of patients with advanced STS are not curative but aim to improve patients' HRQoL through reduction of symptoms, slowing or halting disease progression, and may extend life for some patients. Despite this, there is little research into the impact of chemotherapy on HRQoL for advanced STS patients. In order for patients to make an informed decision about chemotherapy and the predicted effects on all aspects of their lives, clinicians should be able to provide data on HRQoL. This will also enhance the shared decision-making process between clinicians and their patients. Given that survival benefits of treatment beyond 2nd line chemotherapy are marginal, and HRQoL data are lacking for patients treated with third line systemic treatment, simultaneous collection of HRQoL data in patients treated with 1st and 3rd line chemotherapy will enable assessment of the course of HRQoL in patients at the beginning, and further along, their treatment trajectory. After discontinuation of 1st or 3rd line chemotherapy, all patients will be followed up at 2-3 month intervals to determine trajectory of quality of life over time, irrespective of whether or not they receive subsequent line(s) of chemotherapy.

DETAILED DESCRIPTION:
Eligible patients with advanced soft tissue sarcoma will be introduced to this study by their hospital consultant during their routine outpatient appointment. Before deciding if he/she would like to take part, the patient will be provided with a patient information sheet which describes the study in detail. Participation in the study is entirely voluntary and their care will not be affected if he/she chooses not to take part.

The patient information sheet explains that this study involves completing regular questionnaires online, or by paper-and-pencil, about health-related quality of life, expectations of treatment, preferences for making treatment choices and thoughts at the end of chemotherapy.

If a patient agrees to take part, he/she will be asked to sign an informed consent form indicating their willingness to participate. Each patient will be given unique login details to complete the consent form online using the PROFILES website. If he/she prefers to receive paper versions of the questionnaires and complete a paper version of the informed consent form.

After informed consent has been given, each patient will be asked to complete the first questionnaire. This will take around 15-20 minutes to complete. Further questionnaires are completed every time the patient attends hospital for treatment with chemotherapy (each cycle). These questionnaires will take around 10-15 minutes to complete. Most patients have a maximum of six cycles of chemotherapy and therefore will complete six questionnaires during treatment. At the end of chemotherapy, patients will complete one further questionnaire. During follow-up patients will be asked to complete questionnaires online (or by paper) at home every 2-3 months. The maximum time a patient will participate in the study is 2 years.

Only after a participant has given consent, the research team will collect information for their medical files such as the date of their cancer diagnosis and any previous treatments received. This information will be linked to the questionnaire data at the end of the study, in order to analyse whether it is associated with health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of advanced (not amenable to curative surgical resection) soft tissue sarcoma (histology confirmed by sarcoma histopathologist)
* Starting 1st line palliative chemotherapy or 3rd line palliative chemotherapy according to standard treatment guidelines.
* Able to communicate in English
* Mental capacity to provide informed consent and to participate in the study (as determined by the treating physician).
* Patients must be able to complete questionnaires themselves (a prerequisite for 'patient reported outcome' data).
* Patients must be under treatment or follow-up at one of the participating centres

Exclusion Criteria:

* Patients with GIST, Ewing sarcoma, rhabdomyosarcoma and desmoplastic small round cell tumour.
* Patients who have already started 1st line or 3rd chemotherapy.
* Patients who are too ill to receive any further systemic treatment (death is imminent), as determined by the referring health care professional

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years with advanced soft tissue sarcoma.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Change in global health-related quality of life score after treatment with 1st line chemotherapy. | After up to six cycles of chemotherapy (approximately six months)
  Patients will complete the EORTC-QLQ-C30 questionnaire at baseline and each cycle of chemotherapy. Question 30 asks patients to rate their global health-related quality of life on a scale from 1(very poor)- 7 (excellent). After linear transformation, patients will have a score from 0-100. A higher score on global health-related quality of life question means better HRQoL. Change in global HRQoL over treatment with first-line chemotherapy will be presented using descriptive statistics such as mean and standard deviation after each cycle. Change in global HRQoL will be tested using a paired sample t test from baseline to 4 cycles with a 2 sided 5 % significance level. For patients who do not complete 4 cycles, the last score/observation (post baseline) will be carried forward for the analysis.
  A sensitivity analysis will also be performed excluding those patients who do not reach 4 cycles.
  If data is not normally distributed, then the Wilcoxon test will be used.

SECONDARY OUTCOMES:
Change in physical, cognitive, social, role and emotional functioning scores after treatment with first-line chemotherapy. | After up to six cycles of chemotherapy (approximately six months)
  Patients will complete the EORTC-QLQ-C30 questionnaire at baseline and each cycle of chemotherapy. After linear transformation, all functioning scores will produce a score from 0-100. A higher score on the functional scales means better functioning.
Health-related quality of life symptoms scores after treatment with first line chemotherapy | After up to six cycles of chemotherapy (approximately six months)
  Patients will complete the EORTC-QLQ-C30 questionnaire at baseline and each cycle of chemotherapy. After linear transformation, all single items will produce a score from 0-100. A higher score on symptom scales means more complaints.

OTHER OUTCOMES:
Change in global health-related quality of life score after third-line chemotherapy | From start of 3rd line chemotherapy to cessation of 3rd line chemotherapy. (1-12 months)
  Patients will complete the EORTC-QLQ-C30 questionnaire at baseline and each cycle of chemotherapy. Question 30 asks patients to rate their global health-related quality of life on a scale from 1(very poor)- 7 (excellent). After linear transformation, patients will have a score from 0-100. A higher score on global health-related quality of life question means better HRQoL. Change in global HRQoL (continuous) after treatment with third-line chemotherapy will be presented descriptively over time using mean (SD) and graphics.
Patient preference for collaborative decision-making | 2 years.
  Control preference scale: This scale is widely used to measure patient preferences for treatment decision making with health care providers. Patients are asked to chose from five options the phrase that best describes the role that they have
  a) actually taken in dealing with cancer diagnosis/treatment decisions and b) the role that they would have preferred.
  The options are: 1) I prefer to make the final treatment decision. 2) I prefer to make the final treatment decision after seriously considering my doctor's opinion.
  3) I prefer that my doctor and I share responsibility for deciding which treatment is best. 4) I prefer that my doctor makes the final treatment decision, but seriously considers my opinion. 5) I prefer to leave all treatment decisions to my doctor.
  Patients are grouped into those who would prefer an active role in decision making (response 1 or 2), a collaborative role (response 3), or a passive role (response 4 or 5).
Decisional conflict | 2 years
  The decisional conflict scale measures personal perception of decision making and certainty or uncertainty over their choice. This includes determining the level of information and support to make the choice, whether the decision was in line with their values and how satisfied they are, or were, with their decision. Items are given a score value of 0 (no) or 1 (yes). The total score can only be calculated if all four items are answered. The sum of the four items will range from 0 (extremely high decisional conflict) to 4 (no decisional conflict). A score of 3 or less indicates decisional conflict. Results will be descriptive.
Patients' expectations of treatment with chemotherapy | 2 years
  Patients are asked how likely they think that chemotherapy will improve survival, cure their cancer and improve symptoms due to cancer. The answers are on a four point scale: very likely, somewhat likely, a little likely and not likely at all. This single question will enable us to assess expectations of chemotherapy among sarcoma patients and results will be descriptive.
Decisional Regret scores | 2 years
  Patients' retrospective views on their decision to receive chemotherapy will be assessed using the decisional regret scale. Patients are asked to think about the decision they have made and show how strongly they agree/disagree with 5 statements: It was the right decision, I regret the choice that I made, I would go for the same choice if I had to do it over again, the choice did me a lot of harm, the decision was a wise one. Items 2 and 4 should be reverse-coded so that, for each item, a higher number will indicate more regret. To help others interpret the score more readily with other scales ranging from 0 to 100, these scores can then be converted to a 0-100 scale by subtracting 1 from each item then multiply by 25. To obtain a final score, the items are summed and averaged. A score of 0 means no regret; a score of 100 means high regret.
Work ability index scores | 2 years
  The validity and reliability of the work ability has been assessed in correlation analyses and used in many international research studies. These questions assess the ability to work taking into account the demands of the work, health status and resources. There are seven questions from which we selected two general questions to inform future patients who are receiving chemotherapy on their ability to work during and after chemotherapy. These two questions are scored 0-10 and 1-6 will be descriptive scores.
Patient preference for quantity versus quality of life. | 2 years
  Quality-Quantity Questionnaire (QQQ): This tool is a validated construct consisting of eight questions which measure patient attitudes towards tradeoff of quantity versus quality of life (four questions for length of life (LOL) and four questions for quality of life (QOL)). For LOL and QOL a separate score is calculated. The total score for all four questions (LOL or QOL) is calculated and the minimum score (4) is then subtracted. This answer is then divided by the range (20-4) to create a rescaling of 0-100. Decision-making in patients with advanced soft tissue sarcomas is extremely complex. The patients' concerns are of utmost importance when weighing up the benefits and risks of toxic treatment such as chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Winette van der Graaf, PhD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roets E, Younger E, Jones RL, Hollander DD, Azarang L, Desar IME, Young RJ, Oosten AW, de Haan JJ, Gelderblom H, Steeghs N, Husson O, van der Graaf WTA. Health-related quality of life in patients with advanced soft tissue sarcoma receiving first-line palliative chemotherapy (HOLISTIC): longitudinal results from a prospective, observational cohort study. EClinicalMedicine. 2025 Oct 16;89:103561. doi: 10.1016/j.eclinm.2025.103561. eCollection 2025 Nov. PMID 41146924
- [Derived] Younger E, Jones RL, Desar IME, Peckitt C, van der Graaf WTA, Husson O. Health-related quality Of Life In patients with advanced Soft TIssue sarcomas treated with Chemotherapy (The HOLISTIC study): protocol for an international observational cohort study. BMJ Open. 2020 Jun 1;10(6):e035171. doi: 10.1136/bmjopen-2019-035171. PMID 32487574